CLINICAL TRIAL: NCT07335380
Title: Phase IB Trial of Preoperative Lattice-Based Hypofractionated Radiotherapy and Chemo-Immunotherapy for Oral Cavity Squamous Cell Carcinoma
Brief Title: Lattice-Based Radiotherapy and Chemo-Immunotherapy for Oral Cavity Squamous Cell Carcinoma
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: NYU Langone Health (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: 25-00185
Record Dates: First submitted 2026-01-05; First posted 2026-01-13 (Actual); Last update posted 2026-01-29 (Actual); Status verified 2026-01

CONDITIONS: Oral Cavity Squamous Cell Carcinoma
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck | interventions — Drug Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Part 1 - Dose-Escalation (Experimental): Treatment starts at dose level 2 (9 Gy × 3 lattice fractions). A single "sentinel" patient is treated first; if no dose-limiting toxicity (DLT) occurs, the trial continues in fixed three-patient cohorts. The Bayesian Optimal Interval (BOIN) algorithm, set to a target DLT rate of 20%, governs escalation or de-escalation among the three prespecified dose levels (8, 9 and 10 Gy × 3). The principal objective of Part 1 is to identify the maximum tolerated dose (MTD).
  Interventions: Drug: Chemotherapy; Radiation: Lattice Radiotherapy (LRT)
- Part 2 - Expansion (Experimental): All Part 2 subjects receive the MTD together with chemo-immunotherapy.
  Interventions: Drug: Chemotherapy; Radiation: Lattice Radiotherapy (LRT)

INTERVENTIONS:
Drug: Chemotherapy — Patients receive standard induction chemoimmunotherapy (carboplatin, paclitaxel, and pembrolizumab) in three 21-day cycles, beginning on Day 1.
Radiation: Lattice Radiotherapy (LRT) — LRT is administered concurrently with the first cycle of chemoimmunotherapy according to the dose-finding rules

SUMMARY:
Single-arm, two-part, phase IB safety study that uses a Bayesian Optimal Interval (BOIN-12) dose-escalation scheme.

Part 1 (Dose Finding) - Sentinel start at 9 Gy × 3 followed by fixed 3-patient BOIN cohorts exploring 8 Gy × 3 → 9 Gy × 3 → 10 Gy × 3. Target DLT rate θ = 0.20; ≈ 7-15 participants.

Part 2 (Expansion) - Additional enrolment at the selected maximum tolerated dose (MTD) until ≈ 30 evaluable subjects (Parts 1 + 2 combined). Patients receive peaks to the primary tumor alone (Group A) or to the primary + involved nodes (Group B) at the investigators' discretion (non-random).

Surgery occurs 6-8 weeks after RT; adjuvant therapy is pathology-driven.

ELIGIBILITY:
Inclusion Criteria:

* Non-metastatic, pathologically confirmed oral cavity squamous cell carcinoma, cT3-T4a cN0-N3 or cT1-T2 cN1-N3. Histologic variants will be included (papillary squamous cell carcinoma and basaloid squamous cell carcinoma, e.g.). Cytologic diagnosis from a cervical lymph node is sufficient in the presence of clinical evidence of a primary tumor in the oral cavity (oral tongue, floor of mouth, alveolar ridge, buccal or lip, i.e.)
* Surgically resectable
* Zubrod Performance Status of 0-1
* (Phase I) Primary and lymph node ≥ 3 cm
* (Phase II) Primary and lymph node ≥ 3 cm OR Primary ≥ 3 cm
* Patients must provide their personal smoking history prior to registration.
* Negative serum pregnancy test within 14 days prior to registration for women of childbearing potential. Female subjects of childbearing potential and male subjects with female partners of childbearing potential must be willing to avoid pregnancy. Female subjects of childbearing potential who are undergoing RT or who are partners to male subjects in the study should avoid sexual activity or use a highly effective method of birth control during sexual intercourse. Acceptable, highly effective methods of birth control include: intrauterine device (IUD)/intrauterine hormone releasing system (IUS), bilateral tube occlusion, vasectomized partner, combined (estrogen and progesterone containing) or progesterone-only hormonal contraceptives (oral, intravaginal, transdermal, injectable).
* Males who are sexually active with women of childbearing potential must agree to follow instructions for method(s) of contraception (abstinence/protection) for the duration of treatment/study participation.
* The patient must provide study-specific informed consent prior to study entry.
* Adequate renal function within 2 weeks prior to registration
* Adequate hematologic function within 2 weeks prior to registration
* Patients who are HIV positive but who have no prior AIDS-defining illness and have CD4 cells of at least 350/mm3 are eligible. HIV-positive patients must not have multi-drug resistant HIV infection or other concurrent AIDS-defining conditions. Patients must not be sero-positive for Hepatitis B (Hepatitis B surface antigen positive or anti-hepatitis B core antigen positive) or sero-positive for Hepatitis C (anti-Hepatitis C antibody positive). However, patients who are immune to hepatitis B (anti-Hepatitis B surface antibody positive) are eligible (e.g. patients immunized against hepatitis B).

Exclusion Criteria:

* Cancers considered to be primarily located in the oropharynx even if p16 negative
* Carcinoma of the neck of unknown primary site origin (even if p16 negative)
* Distant metastasis or adenopathy below the clavicles;
* Gross total excision of both primary and nodal disease; this includes tonsillectomy, local excision of primary site, and nodal excision that removes all clinically and radiographically evident disease.
* Simultaneous primary cancers or separate bilateral primary tumor sites;
* Prior invasive malignancy (except non-melanomatous skin cancer) unless disease free for a minimum of 1095 days (3 years) (for example, carcinoma in situ of the breast, oral cavity, or cervix are all permissible);
* Prior systemic chemotherapy for the study cancer; note that prior chemotherapy for a different cancer is allowable;
* Prior radiotherapy to the region of the study cancer that would result in overlap of radiation therapy fields;
* Severe, active co-morbidity
* Pregnancy; this exclusion is necessary because the treatment in this study may be significantly teratogenic
* Prior allergic reaction to cisplatin
* Exclusion Criteria for MRI: Normal MRI exclusion criteria will apply, including those on the following list. A standard MRI safety form will be used to identify potential conditions warranting exclusion.

  1. Electrical implants such as cardiac pacemakers or perfusion pumps
  2. Ferromagnetic implants such as aneurysm clips, surgical clips, prostheses, artificial heart, valves with steel parts, metal fragments, shrapnel, bullets, tattoos near the eye, or steel implants
  3. Ferromagnetic objects such as jewelry or metal clips in clothing
  4. Claustrophobia
  5. History of seizures

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2026-04 (Estimated); Primary Completion 2031-03 (Estimated); Study Completion 2031-03 (Estimated)

PRIMARY OUTCOMES:
Maximum tolerated dose (MTD) of pre-operative lattice radiotherapy delivered with chemoimmunotherapy | Up to Year 2
  The BOIN (Bayesian Optimal Interval) algorithm will declare the MTD once a dose has an observed dose-limiting toxicity (DLT) rate compatible with the target toxicity level (θ = 0.20) and all higher doses are ruled out for excess risk.

SECONDARY OUTCOMES:
Percentage of participants with complete pathologic response (pCR) | Up to Year 2
Percentage of participants with major response | Up to Year 2
  Defined as ≤ 10 % viable tumor.
Percentage of participants with macroscopic residual disease | Up to Year 2
  Defined as > 10 % viable tumor.
Progression-free survival (PFS) | Up to Year 2
  Time from Day 1 of protocol therapy to locoregional or distant progression or death, estimated with Kaplan-Meier methods.
Overall survival (OS) | Up to Year 2
  Time from Day 1 of therapy to death from any cause, analyzed with Kaplan-Meier curves
Distant-metastasis-free survival (DMFS) | Up to Year 2
  Time to first distant failure or death.

CONTACTS AND LOCATIONS:
Overall Officials: Colin Hill, MD, Principal Investigator — NYU Langone Health
Locations (1):
- NYU Langone Health, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
The de-identified participant data from the final research dataset will be shared upon reasonable request beginning 9 to 36 months after publication or as required by a condition of awards or supporting agreements, provided the requesting investigator executes a data use agreement with NYU Langone Health. This instance of data sharing will also require separate IRB review as well as review from NYU Langone's Data Sharing Strategy Board (DSSB). Requests should be directed to: colin.hill@nyulangone.org. The protocol and statistical analysis plan will be posted on Clinicaltrials.gov only as required by federal regulation or supporting awards and agreements.
Supporting Information: Study Protocol, SAP
Time Frame: Beginning 9 months and ending 36 months following article publication or as required by a condition of awards and agreements supporting the research.
Access Criteria: The investigator who proposed to use the data will be granted access upon reasonable request. Requests should be directed to colin.hill@nyulangone.org To gain access, data requestors will need to sign a data access agreement. This instance of data sharing will also require separate IRB review as well as review from NYU Langone's DSSB.